CLINICAL TRIAL: NCT06120634
Title: A Quasi-experimental Study Comparing Outcomes and Parent's Responses in 600+ Circumcised Boys in a Lower-Middle Income Country
Brief Title: Comparison of Outcomes of Circumcision Via Open and Plastibell Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehsil Headquarter Hospital (Other Government)
Responsible Party: Principal Investigator, Ali Kamran, Principal investigator, Tehsil Headquarter Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 794/MS/THQ/FW
Record Dates: First submitted 2023-09-25; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Circumcision, Male
Keywords: Circumcision; Open method; Plastibell method; Complications; Outcomes; Parental response

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open surgical method (Active Comparator): In this group, the participants were circumcised using the open method. A total of 304 patients were enrolled in this group.
  Interventions: Procedure: Open surgical method
- Plastibell method (Active Comparator): A total of 304 patients were enrolled in this group and underwent the process of circumcision by the Plastibell method.
  Interventions: Procedure: Plastibell method

INTERVENTIONS:
Procedure: Open surgical method — After separating the preputial skin from glans and removing smegma, two artery clips were applied on the dorsal skin in the center to mark the skin to be divided. Crushing the skin for a couple of minutes, prior to incising, helps to reduce bleeding. The skin was cut about 2-3 mm short of the coronal sulcus. Similarly, 2-3 mm cuff of prepuce was circumferentially cut proximal to the corona. Using bipolar diathermy or catgut 4/0, frenular artery along with dorsal artery and vein of penis were coagulated or ligated respectively to achieve hemostasis. The skin and prepuce were approximated and sutured with catgut 4/0 at four places- ventral, dorsal, and two lateral points. Finally, a dressing with antibiotic ointment was applied to the wound.
  Arms: Open surgical method
Procedure: Plastibell method — The prepuce was separated all around the glans, up to the coronal sulcus, and smegma was removed. A dorsal slit in the skin was made, after crushing the skin for a couple of minutes, long enough to accommodate the passage of an appropriate-sized plastibell. Once the distal edge of the bell snugly fit at or near the coronal sulcus, a ligature was applied and tightened around the sulcus on the bell. The extra preputial skin was cut with either scissors or a surgical blade, after breaking apart and discarding the handle of the plastibell. The urethral meatus was examined and its visibility was ensured prior to returning the baby boy to his parents. The baby was kept under observation for 30 minutes in the surgical ward and re-examined to ensure there was no hematoma or bleeding.
  Arms: Plastibell method

SUMMARY:
Circumcision is considered one of the most common elective surgical procedures, particularly among Muslim and Jewish males. Of all the available techniques, Plastibell is gaining traction amongst surgeons due to its safety in the form of a lower complication rate. The current quasi-experimental study aimed to compare the Open and Plastibell methods of circumcision in a study population which comprised of boys up to 5 years of age who were grouped into the Open method and Plastibell based on parental preference. Follow-up occurred on the 5th, 10th, and, 30th post-procedural day. Basic demographic data, procedural duration, and outcomes were documented.

DETAILED DESCRIPTION:
This study was conducted to compare the Open and Plastibell method of circumcision in boys up to 5-years of age, in terms of procedural time, outcomes and parental satisfaction.

This was a quasi-experimental study of boys up to 5-years of age. Boys meeting the inclusion criteria were categorized into two groups based on parental preference - Open method and Plastibell. Patients were followed-up on the 5th, 10th and 30th post-procedural day. Basic demographic data, procedural duration, and outcomes were documented.

Of 646 boys brought to the hospital for circumcision, 608 met the inclusion criteria with equal participants in both groups. The median age in Open and Plastibell groups was three and five months respectively. The median operating time was significantly shorter in the Plastibell group (4.2 min) compared to the Open method (13 min). Of the complications recorded in 91 children, more were observed in Plastibell group. Post-procedure bleeding occurred in 1.2% children (n=7). Open method resulted in infection, excessive skin removal (n=8 each) and urinary retention (n=7) whereas Plastibell impaction (n=21) and inadequate skin removal (n=19) were the commonest complications in the Plastibell group which were significantly associated with age of the boys. There were no serious adverse events. Open method was preferred by parents for cosmesis and Plastibell for ease of care.

It is concluded that Plastibell, compared to open method, is a quicker method of circumcision and is safe for boys up to 5-years of age, however, earlier circumcisions are associated with lesser complications. The follow-up ensures patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males up to 5 years of age
* Signed, informed consent of parents/guardians

Exclusion Criteria:

* Boys with bleeding disorders, severe jaundice, or genital abnormalities like hypospadias, epispadias, congenital chordee.
* Whose parents did not give consent
* Boys with a larger glans size not feasible for Plastibell circumcision

Ages: 1 Month to 60 Months | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 608 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Post-operative bleeding | From post-operative day 0 to day+30
  Bleeding from the site of circumcision
Post-operative urinary retention | From post-operative day 0 to day+30
  Urinary retention by the patient as reported by the parents/guardians/caregivers
Infection | From post-operative day 0 to day+30
  Swelling, pain, redness, warm to touch as felt by the parents/guardians/caregivers
Over circumcision | From post-operative day 0 to day+30
  Total number of participants with extra skin removed during the circumcision than required
Under circumcision | From post-operative day 0 to day+30
  Number of participants with less skin removed during the circumcision covering half of glans penis
Bell impaction | From post-operative day 0 to day+30
  Number of participants with the head of the penis gets stuck to the Plastibell
Delayed shedding of the ring | From post-operative day 0 to day+10
  Number of participants with failure of Plastibell to shed on its own
Post-procedural phimosis/paraphimosis | From post-operative day 0 to day+30
  Number of participants with entrapment of a retracted foreskin behind the coronal sulcus

SECONDARY OUTCOMES:
Ease of care | From post-operative day 0 to day+30
  total number of Parents' ease in the change of diapers, clothes, and giving bath to the baby assessed subjectively through interview of parents
Satisfaction with cosmetic appearance | From post-operative day 0 to day+30
  Total number of parents satisfied with the appearance of penis after the circumcision

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kamran, FCPS, Principal Investigator — Tehsil Headquarters Hospital Ferozewala, Sheikhupura, Punjab
Locations (1):
- Tehsil Headquarters Hospital Ferozewala, Sheikhupura, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No